CLINICAL TRIAL: NCT01322659
Title: Weaning Using Noninvasive Positive Pressure Ventilation by Means of Helmet in Patients With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1926P
Record Dates: First submitted 2011-03-21; First posted 2011-03-24 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2011-03

CONDITIONS: Inadequate or Impaired Breathing Pattern or Ventilation
Keywords: Mechanical ventilation; Weaning; Noninvasive ventilation; Acute respiratory failure; Helmet
MeSH Terms: conditions — Respiratory Aspiration | interventions — Head Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Helmet NPPV (Active Comparator): Weaning from mechanical ventilation with noninvasive positive pressure ventilation (NPPV)delivered by means of the helmet
  Interventions: Device: Helmet
- ETT IMV (Sham Comparator): Weaning from mechanical ventilation with standard invasive mechanical ventilation (IMV) delivered by means of the endotracheal tube (ETT)
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Helmet — Weaning from mechanical ventilation with noninvasive positive pressure ventilation delivered by means of the helmet
  Arms: Helmet NPPV
Device: Endotracheal tube — Weaning from mechanical ventilation with invasive mechanical ventilation delivered by means of the endotracheal tube
  Arms: ETT IMV

SUMMARY:
The purpose of this study is to determine whether helmet is effective as device for noninvasive positive pressure ventilation in the weaning from mechanical ventilation.

DETAILED DESCRIPTION:
The clinical efficacy of noninvasive positive pressure ventilation (NPPV) has been demonstrated. Interest has emerged in using NPPV to facilitate earlier removal of an endotracheal tube and decrease complications associated with prolonged intubation. Studies assessing NPPV in weaning are not enough and generally are performed with face masks as device for NPPV. This study assesses the efficacy of helmet as device for NPPV during weaning from mechanical ventilation in an ICU and compares this procedure with invasive mechanical complication (IMV) by analyzing respiratory parameters, clinical course and complications.

ELIGIBILITY:
Inclusion Criteria:

* endotracheal mechanical ventilation for 48 hours or more for acute respiratory failure,
* patient ready to be weaned (steady respiratory and hemodynamic conditions for 24 hours),
* spontaneous breathing trial failure
* written informed consent obtained (patient or family)

Exclusion Criteria:

* respiratory and hemodynamic instability
* initial difficult intubation
* bronchial hypersecretion at the weaning time
* non cooperant patient
* recent history of upper gastro-intestinal surgery
* recent history of myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Weaning using noninvasive positive pressure ventilation by means of helmet in patients with acute respiratory failure | 30 days
  Main end-point defined as the weaning success/failure rate

SECONDARY OUTCOMES:
Weaning using noninvasive positive pressure ventilation by means of helmet in patients with acute respiratory failure | 180 days
  * Intubation duration
  * Total duration of mechanical ventilation (endotracheal and non invasive)
  * Weaning process duration
  * Stress response evaluation
  * Daily duration of ventilatory support
  * ICU lentgh of stay
  * Hospital lentgh of stay

CONTACTS AND LOCATIONS:
Overall Officials: Michele Carron, MD, Principal Investigator — University medical hospital of Padova
Locations (1):
- University Medical Hospital, Padua, Italy

REFERENCES:
- [Derived] Carron M, Rossi S, Carollo C, Ori C. Comparison of invasive and noninvasive positive pressure ventilation delivered by means of a helmet for weaning of patients from mechanical ventilation. J Crit Care. 2014 Aug;29(4):580-5. doi: 10.1016/j.jcrc.2014.03.035. Epub 2014 Apr 5. PMID 24793658